CLINICAL TRIAL: NCT07264712
Title: The Effect of Wound Care Education Given to Patients Undergoing Prosthetic Surgery on Wound Care Knowledge, Self-Care Self-Efficacy, and Quality of Recovery
Brief Title: The Effect of Wound Care Education Given to Patients on Wound Care Knowledge, Self-Care Self-Efficacy, and Quality of Recovery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yeliz Sürme, associate professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/419
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Prosthetic Treatment; Wound Care; Education
Keywords: Wound care; Prosthetic surgery; artificial intelligence

STUDY DESIGN:
Intervention Model Description: designed as a randomized controlled experimental
Who Masked: Outcomes Assessor
Masking Description: The person conducting the statistical analyses in the study will be blinded to the experimental groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The purpose of the study will be explained to the individuals in the experimental group using a face-to-face interview technique, and a patient introduction form will be administered by the researcher one day before surgery. The researcher will then provide patients with visual and verbal wound care training using the "Surgical Patient Wound Care Guide," and the educational materials will be provided. To assess the effectiveness of the training, a Knowledge Level Survey consisting of 10 true/false questions will be administered to patients on the third postoperative day. Two weeks after surgery, the Patient Follow-up Form, Self-Care Self-Efficacy Scale, and Quality of Healing Scale will be completed by phone.
  Interventions: Other: artificial intelligence-supported education
- Control Group (No Intervention): The purpose of the study will be explained to the control group members, and a patient introduction form will be administered by the researcher using a face-to-face interview technique one day before surgery. On the third postoperative day, patients will be administered a Knowledge Level Questionnaire consisting of 10 true/false questions. Two weeks after surgery, the patient follow-up form, the Self-Care Self-Efficacy Scale, and the Quality of Recovery Scale will be completed by phone.

INTERVENTIONS:
Other: artificial intelligence-supported education — The purpose of the study will be explained to the individuals in the experimental group using a face-to-face interview technique, and a patient introduction form will be administered by the researcher one day before surgery. The researcher will then provide patients with visual and verbal wound care training using the "Surgical Patient Wound Care Guide," and the educational materials will be provided. To assess the effectiveness of the training, a Knowledge Level Survey consisting of 10 true/false questions will be administered to patients on the third postoperative day. Two weeks after surgery, the Patient Follow-up Form, Self-Care Self-Efficacy Scale, and Quality of Healing Scale will be completed by phone.
  Arms: Intervention group

SUMMARY:
This study will be conducted as a randomized controlled trial to determine the impact of artificial intelligence-assisted wound care training provided to patients undergoing prosthetic surgery on their wound care knowledge, quality of healing, and self-care self-efficacy. It was planned to include 22 individuals in the experimental group and 22 in the control group. However, considering the potential for data loss, the study was planned to be completed with a total of 50 individuals: 25 in the experimental group and 25 in the control group. Patient Identification Form, Patient Follow-up Form, Knowledge Level Questionnaire, Self-Care Self-Efficacy Scale and Quality of Recovery (QoR-15) Scale were used to collect data.

DETAILED DESCRIPTION:
It is crucial to educate patients and their caregivers who have undergone prosthetic surgeries such as TKA and THA about home care before discharge. Therefore, this study will be conducted as a randomized controlled trial to determine the impact of artificial intelligence-assisted wound care training provided to patients undergoing prosthetic surgery on their wound care knowledge, quality of healing, and self-care self-efficacy. The study population will consist of patients hospitalized in the Orthopedics and Traumatology Department of Erciyes University Health Application and Research Center after total hip and knee replacement surgeries, and the sample will consist of patients who meet the inclusion criteria. With 80% power, an effect size of 0.776, and a 95% confidence interval, it was planned to include 22 individuals in the experimental group and 22 in the control group. However, considering the potential for data loss, the study was planned to be completed with a total of 50 individuals: 25 in the experimental group and 25 in the control group. Patient Identification Form, Patient Follow-up Form, Knowledge Level Questionnaire, Self-Care Self-Efficacy Scale and Quality of Recovery (QoR-15) Scale were used to collect data.

Research data will be collected by the researcher between October 2025 and March 2026. The firstly, begins with the patients' hospitalization prior to surgery, and the assignment to either the experimental or control groups will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing total hip or knee replacement surgery
* Those who volunteer to participate in the study
* Those over 18 years of age
* Those who have no communication problems (language, hearing impairment, etc.)

Exclusion Criteria:

* Patients who have developed a surgical site infection
* Illiterate
* Unable to self-care
* Previously had prosthetic surgery will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level | postoperative day 3
  The researcher-created knowledge survey includes 10 true/false questions aimed at measuring the effectiveness of Surgical Patient Wound Care Education provided to patients. Each question will be evaluated out of 10. The lowest possible score is 0, and the highest is 100. Higher scores indicate higher knowledge levels. Expert opinions will be obtained from three faculty members with expertise in the field to assess the adequacy of the survey's content and scope.
Self-Care Self-Efficacy | 15th day after surgery
  The scale originally developed by Yu et al. to determine individuals' self-care self-efficacy levels was modified by Chica-Pérez et al. to assess self-care self-efficacy in older adults with chronic multimorbidity. The scale was designed as a 5-point Likert-type instrument ranging from "1 = I do not trust myself" to "5 = I trust myself a lot." It consists of 10 items in total. In their study, Chica-Pérez et al. reported Cronbach's alpha coefficients as 0.713 for the subscale "Self-Efficacy in Clinical Knowledge-Based Self-Care Behaviors," 0.822 for "Self-Efficacy in Self-Care," 0.881 for "Self-Efficacy in Monitoring Self-Care," and 0.878 for "Self-Efficacy in Self-Care Management." Chica-Pérez et al. stated that the minimum possible score is 10 and the maximum is 50, with higher scores indicating higher levels of self-efficacy in self-care.
Quality of Recovery | 15th day after surgery
  The Quality of Recovery-15 (QoR-15) is a brief postoperative recovery scale developed and validated by Stark et al. in 2013. It is a shortened version of the QoR-40 scale. It is easier to use because it is shorter and can be completed in a shorter time. Like the QoR-40, it contains 15 questions that assess the patient's pain, physical comfort, physical independence, psychological support, and emotional state. The test results in a score between 0 and 150, with a higher score indicating better recovery quality. With the latest update, the minimal clinically important difference, that is, the lowest difference indicating a meaningful change, is 6 for the QoR-15.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz SÜRME, ASSOCIATE, Principal Investigator — TC Erciyes University
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University, Kayseri, Melikgazi
  - Health training and research hospital, Kayseri, Melikgazi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yıldız GN. Öz bakım öz yeterlilik ölçeği'nin Türkçe geçerlik güvenirliğinin sağlanması: Metodolojik bir araştırma. Turkiye Klinikleri J Nurs Sci, 2025;17(1), 174-183. https://doi.org/10.5336/nurses.2024-105063
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Chica-Perez A, Dobarrio-Sanz I, Correa-Casado M, Fernandez-Sola C, Ruiz-Fernandez MD, Hernandez-Padilla JM. Spanish version of the self-care self-efficacy scale: A validation study in community-dwelling older adults with chronic multimorbidity. Geriatr Nurs. 2023 Sep-Oct;53:181-190. doi: 10.1016/j.gerinurse.2023.07.016. Epub 2023 Aug 2. PMID 37540914
- [Background] Yu DS, De Maria M, Barbaranelli C, Vellone E, Matarese M, Ausili D, Rejane RE, Osokpo OH, Riegel B. Cross-cultural applicability of the Self-Care Self-Efficacy Scale in a multi-national study. J Adv Nurs. 2021 Feb;77(2):681-692. doi: 10.1111/jan.14617. Epub 2020 Dec 9. PMID 33295675
- [Background] Ismail EA, Elshafie MA. Patient-reported outcomes after femoral nerve block versus periarticular injections in patients undergoing total knee arthroplasty: A randomized controlled study. Journal of Cleaner Production, 2021;277(12):123958 https://doi.org/10.1016/j.jclepro.2020.123958